CLINICAL TRIAL: NCT00323817
Title: To Evaluate the Efficacy and Safety in Subjects With Functional Dyspepsia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zeria Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 99010206E
Record Dates: First submitted 2006-05-08; First posted 2006-05-10 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — Z 338

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Z-338

SUMMARY:
To evaluate the efficacy and safety of Z-338 in subjects with Functional Dyspepsia

ELIGIBILITY:
Inclusion Criteria:

* Subjects presenting diagnosis of FD as defined by the Rome II
* Subjects presenting postprandial fullness and/or Early satiety should be the most bothersome symptom

Exclusion Criteria:

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Estimated)
Dates: Start 2006-04; Primary Completion 2009-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Global subject Outcome Assessment | 12 month

SECONDARY OUTCOMES:
Individual symptom | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, PhD, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- Leuven University, Leuven, Belgium